CLINICAL TRIAL: NCT01939249
Title: BIOTRONIK-A Prospective, Randomized, Multicenter Study to Assess the Safety and Effectiveness of the Orsiro Sirolimus Eluting Stent in the Treatment of Subjects With up to Two de Novo Coronary Artery Lesions - IV
Brief Title: Prospective, Randomized, Multicenter Study to Assess the Safety and Effectiveness of the Orsiro Sirolimus-eluting Stent
Acronym: BIOFLOW-IV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Biotronik AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C1204
Record Dates: First submitted 2013-09-06; First posted 2013-09-11 (Estimated); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Abbott Laboratories Xience (Active Comparator): Subjects assigned to Abbott Laboratories Xience can be treated with either the Xience Prime or Xience Xpedition drug eluting stent (DES).
  Interventions: Device: Abbott Laboratories Xience
- Biotronik Orsiro (Experimental): Subjects assigned to Biotronik Orsiro will be treated with Biotronik Orsiro
  Interventions: Device: Biotronik Orsiro

INTERVENTIONS:
Device: Abbott Laboratories Xience
  Arms: Abbott Laboratories Xience
Device: Biotronik Orsiro
  Arms: Biotronik Orsiro

SUMMARY:
BIOFLOW-IV is a prospective, international, multicenter, randomised controlled trial. The purpose of this trial is to compare the Biotronik Orsiro drug eluting stent system with the Xience Prime / Xience Xpedition (Xience)drug eluting stent system in de novo coronary lesions. The study is powered for non-inferiority with respect to Target Vessel Failure(TVF)at 12 months.

ELIGIBILITY:
Main Inclusion Criteria:

* Subject must provide written informed consent
* The target reference vessel diameter (RVD) is ≥ 2.50 mm and ≤ 3.75 mm assessed either visually or by online QCA.
* Target lesion length is ≤ 26 mm (assessed either visual estimate or by online QCA) and can be covered by one study stent
* Single de novo lesion with ≥ 50% and < 100% stenosis in up to 2 coronary arteries

Main Exclusion Criteria:

* Subject has evidence of myocardial infarction within 72 hours prior to the index procedure
* Planned intervention of non-target vessel(s) within 30 days after the index procedure
* Planned intervention of target vessel(s) after the index procedure
* Target lesion is located in the left main
* Target lesion is located in or supplied by an arterial or venous bypass graft
* Target lesion involves a side branch > 2.0 mm in diameter by visual estimate or by online QCA
* Proximal or distal to the target lesion located stenosis that might require future revascularization or impede run off

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 585 (Estimated)
Dates: Start 2013-09; Primary Completion 2016-03-23 (Actual); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Target Vessel Failure | 12 months post index procedure

SECONDARY OUTCOMES:
Rate of clinically-driven target lesion revascularization (TLR) | 1-month, 6-month, 12-month, 2-year, 3-year, 4-year and 5-year
Rate of clinically-driven target vessel revascularization (TVR) | 1-month, 6-month, 12-month, 2-year, 3-year, 4-year and 5-year
Rate of target lesion failure (TLF), defined as composite of cardiac death, target vessel Q-wave or non-Q wave myocardial infarction (MI), emergent coronary artery bypass graft (CABG), any clinically-driven TLR | 1-month, 6-month, 12-month, 2-year, 3-year, 4-year and 5-year

CONTACTS AND LOCATIONS:
Overall Officials: Shigeru Saito, MD, Principal Investigator — Okinawa Tokushukai Shonan Kamakura General Hospital; Ton Slagboom, MD, Principal Investigator — Onze Lieve Vrouwe Gasthuis
Locations (45):
- Australia (2):
  - Fiona Stanley Hospital, Murdoch
  - Prince of Wales Hospital Sydney, Sydney
- Belgium (2):
  - Gasthuisberg Leuven, Leuven
  - AZ Delta, H. Hart Roeselare, Roeselare
- Roskilde Sygehus Nord, Roskilde, Denmark
- Germany (8):
  - Universitäts-Herzzentrum Freiburg Bad Krozingen, Bad Krozingen
  - Herz- und Diabeteszentrum NRW - Kardiologische Klinik, Bad Oeynhausen
  - Segeberger Kliniken GmbH, Bad Segeberg
  - Charite Campus Mitte - Med. klinik für Kardiologie, Berlin
  - Universitätsklinik Bonn, Bonn
  - Amper Kliniken AG, Dachau
  - Medizinische Hochschule Hannover (MHH), Klinik für Kardiologie und Angiologie, Hanover
  - Medizinische Klinik 8-Kardiologie -Klinikum Nürnberg Sued, Nuremberg
- Israel (3):
  - Rambam Health Corporation, Rambam Medical Center, Batgalim, Haifa
  - Hedasit Medical Research Services and Development Ltd. Hadassah Ein-Kerem Medical Center Kiryat Hadassah, Jerusalem
  - Clalit Health Services, Rabin Medical Center, Cardiology, Petah Tikva
- Japan (11):
  - Tenjinkai Shinkoga Hospital, Fukuoka
  - Akanekai Tsuchiya General Hospital, Hiroshima
  - Hospital Hakodate, Hokkaido
  - Sakurakai Takahashi Hospital, Hyōgo
  - Japan Organization of Occupational Health and Safety Kanto Rosai Hos-pital, Kanagawa
  - Okinawa Tokushukai Shonan Kamakura General Hospital, Kanagawa
  - Saiseikai Yokohamashi Tobu Hospital, Kanagawa
  - Japan Organization of Occupational Health and Safety Kansai Rosai Hospital, Kumamoto
  - Japan Organization of Occupational Health and Safety Kumamoto Rosai Hospital, Kumamoto
  - Toho University Ohashi Medical Center, Tokyo
  - Tokai University Hachioji Hospital, Tokyo
- Netherlands (4):
  - Onze Lieve Vrouwe Gasthuis (OLVG), Amsterdam
  - Tergooi Blaricum, Blaricum
  - Amphia Hospital, Breda
  - Isala Klinieken, Zwolle
- Cardiology Department, Christchurch Hospital, Christchurch, New Zealand
- Poland (4):
  - University Hospital Krakow, Krakow
  - Miedziowe Centrum Zdrowia SA, Lubin
  - Clinical Hospital Medical University Poznan, Poznan
  - General Cardiology & Haemodynamics Dept., Institute of Cardiology, Warsaw
- Spain (4):
  - Hospital del Mar, Barcelona
  - Hospital Clínico y Provincial de Barcelona, Barcelona
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Virgen de la Macarena, Seville
- Sweden (2):
  - Universitetssjukhuset Örebro, Oerebrö
  - Akademiska Sjukhuset, Uppsala
- Switzerland (3):
  - University Hospital Lausanne, Lausanne
  - CardioCentro Ticino, Lugano
  - University Hospital Zürich, Zurich

REFERENCES:
- [Derived] Mankerious N, Toelg R, Abdelghani M, Garcia-Garcia HM, Farhan S, Allali A, Windecker S, Lefevre T, Saito S, Kandzari DE, Waksman R, Richardt G, Hemetsberger R. Impact of coronary artery tortuosity on outcomes following stenting with newer-generation drug-eluting stents. An analysis of the randomized BIOFLOW trials. Rev Esp Cardiol (Engl Ed). 2025 Aug;78(8):682-691. doi: 10.1016/j.rec.2024.12.009. Epub 2025 Jan 4. English, Spanish. PMID 39761745
- [Derived] Hemetsberger R, Mankerious N, Toelg R, Abdelghani M, Farhan S, Garcia-Garica HM, Allali A, Windecker S, Lefevre T, Saito S, Kandzari D, Waksman R, Richardt G. Patients with higher-atherothrombotic risk vs. lower-atherothrombotic risk undergoing coronary intervention with newer-generation drug-eluting stents: an analysis from the randomized BIOFLOW trials. Clin Res Cardiol. 2023 Sep;112(9):1278-1287. doi: 10.1007/s00392-023-02205-4. Epub 2023 Apr 16. PMID 37062047
- [Derived] Hemetsberger R, Abdelghani M, Toelg R, Garcia-Garcia HM, Farhan S, Mankerious N, Elbasha K, Allali A, Windecker S, Lefevre T, Saito S, Kandzari D, Waksman R, Richardt G. Complex vs. non-complex percutaneous coronary intervention with newer-generation drug-eluting stents: an analysis from the randomized BIOFLOW trials. Clin Res Cardiol. 2022 Jul;111(7):795-805. doi: 10.1007/s00392-022-01994-4. Epub 2022 Feb 25. PMID 35212802
- [Derived] Hemetsberger R, Abdelghani M, Toelg R, Mankerious N, Allali A, Garcia-Garcia HM, Windecker S, Lefevre T, Saito S, Slagboom T, Kandzari D, Koolen J, Waksman R, Richardt G. Impact of Coronary Calcification on Clinical Outcomes After Implantation of Newer-Generation Drug-Eluting Stents. J Am Heart Assoc. 2021 Jun 15;10(12):e019815. doi: 10.1161/JAHA.120.019815. Epub 2021 May 29. PMID 34056911
- [Derived] Dan K, Garcia-Garcia HM, Kolm P, Windecker S, Saito S, Kandzari DE, Waksman R. Comparison of Ultrathin, Bioresorbable-Polymer Sirolimus-Eluting Stents and Thin, Durable-Polymer Everolimus-Eluting Stents in Calcified or Small Vessel Lesions. Circ Cardiovasc Interv. 2020 Sep;13(9):e009189. doi: 10.1161/CIRCINTERVENTIONS.120.009189. Epub 2020 Sep 8. PMID 32895004
- [Derived] Toelg R, Slagboom T, Waltenberger J, Lefevre T, Saito S, Kandzari DE, Koolen J, Richardt G. Individual patient data analysis of the BIOFLOW study program comparing safety and efficacy of a bioresorbable polymer sirolimus eluting stent to a durable polymer everolimus eluting stent. Catheter Cardiovasc Interv. 2021 Nov 1;98(5):848-856. doi: 10.1002/ccd.29254. Epub 2020 Sep 5. PMID 32890442
- [Derived] Saito S, Toelg R, Witzenbichler B, Haude M, Masotti M, Salmeron R, Witkowski A, Uematsu M, Takahashi A, Waksman R, Slagboom T. BIOFLOW-IV, a randomised, intercontinental, multicentre study to assess the safety and effectiveness of the Orsiro sirolimus-eluting stent in the treatment of subjects with de novo coronary artery lesions: primary outcome target vessel failure at 12 months. EuroIntervention. 2019 Dec 6;15(11):e1006-e1013. doi: 10.4244/EIJ-D-18-01214. PMID 31235458